CLINICAL TRIAL: NCT00220844
Title: Effect of Tricyclic Antidepressant Agents on Gastric Accommodation and Emptying
Brief Title: Tricyclic Antidepressants (TCAs) on Gastric Emptying
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Futility; study coordinator left and were unable to continue data collection; missing data
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TU4255
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Dyspepsia
MeSH Terms: conditions — Dyspepsia | interventions — Desipramine; Amitriptyline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nortriptyline (Experimental)
  Interventions: Drug: Desipramine
- Placebo (Experimental)
  Interventions: Drug: Amitriptyline

INTERVENTIONS:
Drug: Desipramine
  Arms: Nortriptyline
Drug: Amitriptyline
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effects of two tricyclic antidepressant agents (TCAs), amitriptyline and desipramine, on gastric emptying and gastric accommodation using a newly developed scintigraphic test that simultaneously measures both gastric emptying and gastric volume (accommodation). These two tricyclic antidepressant agents are commonly used at low doses to treat patients with refractory functional dyspepsia.

DETAILED DESCRIPTION:
The normal control subjects will be randomized to receive either amitriptyline or desipramine as the tricyclic antidepressant agent, with 30 subjects per group. Subjects will undergo two outpatient gastric emptying/volume tests and two satiety tests; one of each after 7 days of treatment with oral consumption of the study agent and the other one of each after 7 days of treatment with placebo. The order of the treatments (active drug or placebo) will be randomized with 7 days washout between the studies. During the study, the subjects will consume their regular diet. Subjects will also be randomized to receive either amitriptyline 25 mg po qhs as the active drug or desipramine 25 mg po qhs as the active drug. Side effects of the agents will be monitored during the study.

Each subject will undergo a brief history and physical exam prior to entering the study. The subject will have height and weight measured. A questionnaire will be administered to the subject inquiring about gastrointestinal symptoms and medical history. This is to screen for a history of underlying pulmonary, cardiovascular, or gastrointestinal disease. Females will be studied only during the follicular phase (days 1-10) of the menstrual cycle, to minimize the effect of the menstrual cycle on motility (Wald, at al). In addition, females will be given pregnancy screening with a urine beta-human chorionic gonadotropin pregnancy test (Sure-Vue; Fisher Scientific, Inc) prior to the start of the study.

For the simultaneous gastric volume/emptying tests, subjects will be studied in the fasting condition. The study subject history and physical examination form will be filled out which captures information on symptoms for the last week. An intravenous line will be started. The subject will take study medication with a small sip of water. After 10 minutes, 10 mCi 99mTc pertechnetate will be infused intravenously over 30 seconds. Imaging of the stomach will be performed with a gamma camera 20 minutes after injection with both anterior and posterior imaging followed by SPECT imaging using the General Electric Dual Head MAXXUS (General Electric Medical Systems) connected to a General Electric Starcam 4000i computer. A total of 360o rotation around the subject will be obtained using a circular orbit (32 stops at 15 sec per stop) with the heads for the camera close to the subject. After this, the patient will ingest an egg sandwich labeled with 300 µCi 111Indium-oxine cooked into the eggs to label the solid material. The subject will consume 300 ml of unlabelled water. Imaging will then commence immediately after meal ingestion (time 0) for 111In counts to assess solid-phase gastric emptying using both anterior and posterior imaging. This will be followed immediately by imaging for the 99mTc counts to assess gastric volumes. Imaging for 99mTc will be performed with SPECT 3-D imaging. These will be repeated at 20, 40, 60, 80, 100, 120, 150, 180, 210, and 240 minutes after the meal ingestion. Our prior studies show that 4 hour gastric emptying best characterizes gastric emptying. Peak gastric accommodation occurs at 0-40 minutes. At the time of each imaging, symptoms will be monitored. Symptoms of abdominal fullness, nausea, abdominal discomfort, and bloating will be graded by the study subject from 0 (none) to 5 (severe). In addition, an inquiry into possible side effects to TCAs (sedation, confusion, disturbed concentration, dry mouth, constipation, nausea, and urinary retention) will be made.

On the next day, the subject will return in a fasting condition for the satiety test. The methods are similar to those of Tack et al and Chial et al. The subject will take their study medication. After 30 minutes, the subject will drink the nutrient drink Ensure at a rate of 100 ml every 5 minutes until the subject feels completely full. After each 100 ml, symptoms will be monitored, scoring the symptoms of satiety (fullness), nausea, abdominal discomfort, and bloating on a scale of (0-5). The volume of Ensure consumed by the subject will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Sixty normal subjects, males and females within the ages of 18 to 65 years, will be studied. Normal control subjects will be recruited for voluntary participation through poster advertisements. A normal subject is defined as a person with no gastrointestinal (GI) symptoms; no prior history of peptic ulcer disease or irritable bowel disease; no previous history of a GI motility disorder (including, but not limited to, achalasia, gastroparesis); on no medications for GI disorders; no history of prior surgery on the GI tract (esophagus, stomach, large or small intestine); and a normal physical examination.

Exclusion Criteria:

* History of a motility disorder (including, but not limited to, achalasia, gastroparesis)
* History of peptic ulcer disease
* Symptoms referable to gastric dysmotility (nausea, vomiting, early satiety, heartburn, postprandial abdominal distension)
* Use of medications that may affect GI motor function (beta adrenergic receptor blockers, calcium channel blockers, histamine type 2 receptor antagonists, proton pump inhibitors, prokinetic agents, antidepressants, and the use of narcotic analgesics)
* Regular use of nonsteroidal anti-inflammatory medications
* Use of monoamine oxidase inhibitors
* Pregnancy or breast feeding
* Prior gastrointestinal surgery (except appendectomy)
* Contraindications to amitriptyline or desipramine, which will be exclusion criteria to the study, include hypersensitivity or allergy to any tricyclic drug, concomitant therapy with a monoamine oxidase inhibitor, recent myocardial infarction, myelography within previous 48 hours, or lactation. In addition, history of prostate problems, history of urinary retention, known glaucoma, history of seizures, or thyroid or liver dysfunction are exclusionary criteria to the use of TCAs and to entry into this study.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Gastric emptying | 4 hours
Gastric volume | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Henry P Parkman, MD, Principal Investigator — Temple University
Locations (1):
- Temple University School of Medicine, Philadelphia, Pennsylvania, United States